CLINICAL TRIAL: NCT02613390
Title: A Pilot Study to Evaluate Safety of Intraoperative MRI-Based Image Guidance for Laser Ablation of Epidural Metastasis
Brief Title: Safety Evaluation of Intra-Operative MRI-Based Guidance for Laser Ablation of Epidural Metastasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2015-0481; NCI-2015-02277 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2015-11-20; First posted 2015-11-24 (Estimated); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Spinal Tumor
Keywords: Epidural metastasis; Magnetic resonance imaging; MRI; Guidance system; Spinal surgery; Questionnaires; Surveys
MeSH Terms: conditions — Spinal Cord Neoplasms | interventions — Magnetic Resonance Spectroscopy; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRI-Based Image Guidance (Experimental): MRI images of the spine taken of anesthetized participant in the operative prone position. These images are exported into a computer navigation program, and used to help the doctor perform surgery.
  Pain and symptom questionnaires completed at baseline and at follow up.
  Interventions: Procedure: Magnetic Resonance Imaging (MRI); Behavioral: Questionnaires

INTERVENTIONS:
Procedure: Magnetic Resonance Imaging (MRI) — MRI images of the spine taken of anesthetized participant in the operative prone position.
  Other Names: MRI
Behavioral: Questionnaires — Pain and symptom questionnaires completed at baseline and at follow up.
  Other Names: Surveys

SUMMARY:
The goal of this clinical research study is to learn about the safety and accuracy of using MRI as a guidance system during laser ablation surgery of tumors that have spread to the spine.

DETAILED DESCRIPTION:
Study Visits:

If you agree to take part in this study, before your surgery:

* You will have a physical exam.
* You will have a neurological exam (tests to check the functioning of your nerves, including tests of your balance and reflexes).
* You will complete questionnaires about pain and other symptoms that should take about 10-15 minutes.
* You will sign a separate consent for your spinal surgery that explains the risks.

During the Surgery:

You will be positioned lying face down on your stomach during surgery. While you are under anesthesia, an MRI will be used to take images of your spine. This is an intraoperative MRI, meaning that it is performed in a special magnet located inside a specifically designed operating room. These images will be loaded into a computer navigation program and will be used to help the doctor perform surgery.

Markers will also be attached to the skin of your back. These markers are used together with the navigation program and MRI images to record the location of where on your spine the doctor should cut. This recording will be compared to the MRI images.

Your doctor will check the accuracy of this recording in 2 ways:

* Placing the tip of the navigation probe on your skin and comparing it with the computer calculation in the computer navigation program. This is a standard navigation probe commonly used in spinal surgeries.
* Inserting the navigation probe through a small cut on your skin along the surgical area and taking an x-ray image of its location.

If there is a difference in the result of these 2 measurements, your doctor will use the result of the first step to check the accuracy of the MRI image.

If there is more than 2 millimeter difference between the visual inspection position and the computer model position, your doctor may decide to do one of the following steps:

* Restart the recording process by getting a new MRI image
* Use only the x-ray images to complete the procedure
* Stop the surgery

On the Day After Surgery:

* You will have a physical exam.
* You will have a neurological exam.
* You will complete the same questionnaires as before.

Follow-Up Visits:

The research staff will call you 3 weeks after surgery to ask about your recovery and you will be asked to answer the same questionnaires as before.

You will return for a follow-up visit after surgery:

* You will have a physical exam.
* You will have a neurological exam.
* You will complete the same questionnaires as before.

Length of Study Participation:

Your participation in the study will be over after your follow-up visit.

You will be taken off study if during surgery the doctor thinks the navigation is not accurate, you are injured related to an inaccurate image guidance, or your surgery is stopped.

This is an investigational study. The MRIs and x-rays on this study are performed using FDA-approved and commercially available methods. The use of MRI as image guidance for spinal surgery is investigational.

Up to 10 participants will be enrolled in this study. All will take part at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Age =/> 18 years old.
2. Must have epidural metastasis to be treated with MRI-guided laser ablation.
3. Vertebral body site to be treated is located from C3 to L5.
4. Signed informed consent.

Exclusion Criteria:

1. Requires open spinal procedure or a percutaneous procedure without the use of image guidance.
2. Unable to tolerate general anesthesia and prone position.
3. Unable to undergo MRI of the spine.
4. Pregnant female.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-12-18 (Actual); Primary Completion 2018-10-17 (Actual); Study Completion 2018-10-17 (Actual)

PRIMARY OUTCOMES:
Safety determined by 0% frequency of intraoperative and perioperative adverse events | 3 weeks
  Safety of Intraoperative MRI-Based Image Guidance to Perform Laser Ablation of Epidural Metastasis

SECONDARY OUTCOMES:
Accuracy of MRI-Based Image Guidance to Perform Laser Ablation of Epidural Metastasis | 1 day
  Navigation considered inaccurate if there is a discrepancy of more than 2mm between the real position of the probe confirmed by direct visual inspection, and the computer model displayed on the navigation screen.

CONTACTS AND LOCATIONS:
Overall Officials: Claudio E. Tatsui, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org